CLINICAL TRIAL: NCT02735174
Title: Phase 4: Improving Asthma Outcomes By Facilitating Patient-Centered Care At School (Asthma-Free School)
Brief Title: Improving Asthma Care by Partnering With School Nurses to Bring Asthma Care Into the Inner-City Schools
Acronym: AFS4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Verizon Foundation (Other); Luther Foundation (Other)
Responsible Party: Principal Investigator, Theresa Guilbert, MD, M.D., Professor Division of Pulmonary Medicine, Children's Hospital Medical Center, Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIN001_AFS4
Record Dates: First submitted 2016-02-17; First posted 2016-04-12 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Asthma
Keywords: Telehealth; Sensor cap; School based care; Community health; AsthmaTreatSmart Application
MeSH Terms: conditions — Asthma | interventions — Nebulizers and Vaporizers; Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm asthma self-management (Experimental): Interventions include:
  Sensor cap system for inhalers App for SmartPhone Motivational interviews Telehealth clinic visits
  Interventions: Device: Sensor cap system for inhalers; Other: App for SmartPhone; Behavioral: Motivational interviews; Other: Telehealth clinic visits

INTERVENTIONS:
Device: Sensor cap system for inhalers — All subjects will be given a commercially available inhaler cap with monitoring sensor on clinically prescribed asthma inhalers.
  Other Names: Propeller
Other: App for SmartPhone — All subjects will be given smart phone with mobile software management platform to motivate and record medication adherence.
Behavioral: Motivational interviews — All subjects will have motivational telehealth visits to assess adherence and promote problem-solving skills
Other: Telehealth clinic visits — All subjects will have asthma medical visits via telehealth technology to assess asthma control.

SUMMARY:
This is a pilot study to improve the partnership between Cincinnati Children's Medical Center (CCHMC), Cincinnati Public Schools (CPS), and Cincinnati Health Department (CHD) to reduce childhood asthma in the inner city schools of Cincinnati and CCHMC. We are calling this project "asthma-free schools" and bringing it to neighborhoods where the incidence of asthma is especially high. We have designed this study to work with school-based asthma care programs. Children with high-risk asthma will be asked to participate. "High-risk" will be defined as poorly controlled asthma, frequent school absences, and/or need for daily controller asthma medications. We will use a commercially available inhaler cap sensor to help track medication use and symptoms through a smartphone. The study visits will be done mostly at the school using telehealth technology similar to Skype.

DETAILED DESCRIPTION:
This study is part of a community health collaboration between Cincinnati Children's Hospital Medical Center (CCHMC), the local public health department and designated inner city schools. The purpose is to address school-based asthma care barriers and then to test the efficacy of this program in a pilot study to improve asthma outcomes in 30 urban core youth.

Greater Cincinnati's geography places it at the environmentally tricky confluence of low-lying smog-trapping hills, three heavily traveled interstate highways, and high rate of allergen exposure. This makes it an area ripe for asthma. The overall rate of pediatric asthma in Greater Cincinnati is more than twice the national average and, in some urban-core neighborhoods, as high as 10 times the national rate.

Poor asthma control across the nation and locally in Cincinnati is associated with an overrepresentation of children from minority groups, low-income families, and single parent households who deal with economic hardship and familial strain compared to those with well-controlled asthma. Data show that no more than 50% of patients keep appointments or fill prescriptions, leading to continued poor asthma control and risk for future exacerbation.

This is an interventional pilot study where about 30 high-risk asthmatic participants will be identified to participate and a number of interventions will be incorporated including asthma specific questionnaires, use of a commercially available inhaler cap with monitoring sensor, a mobile software management platform that tracks adherence of all asthma medications, mobile based telehealth medical visits to assess asthma control, and mobile based telehealth adherence problem-solving interventions.

This proposal is funded through a Luther Foundation and Verizon Foundation philanthropic gifts.

ELIGIBILITY:
Inclusion Criteria:

* history of provider diagnosed asthma
* history of uncontrolled asthma in the past 12 months as measured by two asthma control Test (ACT) scores less than 20; or more than or equal to 1 emergency room visit or hospitalization for asthma; or more than or equal to 2 prednisone bursts with current persistent asthma as defined by National Asthma Education and Prevention Program (NAEPP) guidelines
* attendance at participating school

Exclusion Criteria:

* active chronic disease apart from asthma or allergic disease
* plans to change schools during the school year

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2016-01; Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Guilbert, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Asthma Self-management: Interventions include:
  Sensor cap system for inhalers App for SmartPhone Motivational interviews Telehealth clinic visits
  Sensor cap system for inhalers: All subjects will be given a commercially available inhaler cap with monitoring sensor on clinically prescribed asthma inhalers.
  App for SmartPhone: All subjects will be given smart phone with mobile software management platform to motivate and record medication adherence.
  Motivational interviews: All subjects will have motivational telehealth visits to assess adherence and promote problem-solving skills
  Telehealth clinic visits: All subjects will have asthma medical visits via telehealth technology to assess asthma control.
Period: Overall Study
Arm/Group | Single Arm Asthma Self-management
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Asthma Self-management
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.67 (2.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21
Baseline CASI score [Mean (Standard Deviation); unit: score on a scale] — Composite Asthma Severity Index (CASI) score, minimum value 0 and maximum value 20. A lower score shows improvement.
  score on a scale | 4.67 (3.07)

OUTCOME MEASURES:

1. Primary Outcome: Change in Composite Asthma Severity Index (CASI) Score
Description: Change in composite asthma severity index score (Baseline CASI score-6 month CASI score). A positive score indicates a better outcome.
  [The CASI score has a minimum value = 0, maximum value = 20]. The rows represent the change from baseline in scores in all subjects and subsets of participants who obtained "CASI >=4 at baseline and "CASI <4" at baseline.
Time Frame: Baseline to 6 months
Population: 21 participants were analyzed for the CASI score all participants value. Participants were grouped in two categories. 11 participants with baseline CASI >=4 were analyzed independently for the CASI score >=4 at Baseline Value. 10 participants with baseline CASI <4 were also analyzed independently for the CASI score <4 at Baseline Value.
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Single Arm Asthma Self-management
Number analyzed (Participants) | 21
Change in score on a scale
  Change in CASI score all participants | 0.14 (2.90)
  Change in CASI score >=4 at Baseline: number analyzed (Participants) | 11
  Change in CASI score >=4 at Baseline | 2.4 (2.50)
  Change in CASI score <4 at Baseline: number analyzed (Participants) | 10
  Change in CASI score <4 at Baseline | -1.91 (1.22)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Single Arm Asthma Self-management
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT02735174/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT02735174/ICF_001.pdf